CLINICAL TRIAL: NCT03022825
Title: QUILT-3.032: A Multicenter Clinical Trial of Intravesical Bacillus Calmette-Guerin (BCG) in Combination With ALT-803 (N-803) in Patients With BCG Unresponsive High Grade Non-Muscle Invasive Bladder Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-ALT-803-01-16
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Bladder Cancer
Keywords: BCG; bladder cancer; immunotherapy; interleukin-15; intravesical; non-muscle invasive; NMIBC
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BCG+N-803 (Experimental)
  Interventions: Drug: N-803 and BCG; Drug: N-803

INTERVENTIONS:
Drug: N-803 and BCG — BCG and N-803 will be mixed together (with saline) and administered via intravesical instillation weekly for 6 consecutive weeks (induction). After the first disease assessment, eligible patients will receive either a 3-week maintenance course or a 6-week re-induction course (second treatment period) at Month 3. Eligible patients will continue to receive maintenance treatment in the third treatment period at Months 6, 9, 12, and 18. Eligible patients have the option to receive maintenance treatment in the fourth treatment period at Months 24, 30, and 36.
Drug: N-803 — N-803 will be administered via intravesical instillation weekly for 6 consecutive weeks (induction). After the first disease assessment, eligible patients will receive either a 3-week maintenance course or a 6-week re-induction course (second treatment period) at Month 3. Eligible patients will continue to receive maintenance treatment in the third treatment period at Months 6, 9, 12, and 18. Eligible patients have the option to receive maintenance treatment in the fourth treatment period at Months 24, 30, and 36.

SUMMARY:
This is a Phase II/III, open-label, single-arm, multicenter study of intravesical BCG plus N-803 or N-803 only in patients with BCG unresponsive high grade non-muscle invasive bladder cancer (NMIBC). All patients treated in the study will receive via a urinary catheter in the bladder, BCG plus N-803 or N-803 only weekly for 6 consecutive weeks (initial induction treatment period). After the first disease assessment, eligible patients will receive either a 3-week maintenance course or a 6-week re-induction course (second treatment period) at Month 3. Eligible patients will continue to receive maintenance treatment in the third treatment period at Months 6, 9, 12, and 18. Eligible patients have the option to receive maintenance treatment in the fourth treatment period at Months 24, 30, and 36. The study duration is 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age or older
* Histologic confirmation of non-muscle invasive bladder cancer of the transitional cell carcinoma high-grade subtype (mixed histology tumors allowed if transitional cell histology is predominant histology).
* Histologically confirmed presence of BCG-unresponsive CIS (with or without Ta or T1 disease) or histologically confirmed presence of BCG-unresponsive high-grade Ta or T1 disease.
* Absence of resectable disease after transurethral resection (TURBT) procedures (residual carcinoma in situ (CIS) acceptable; patients with T1 tumors must undergo repeat resection and biopsy [inclusive of muscularis propria] if initial biopsy did not include muscularis propria). Patients with high-grade Ta and/or T1 disease should have complete resection before study treatment.
* BCG-unresponsive disease as defined as: (a) Persistent or recurrent CIS (+/- recurrent Ta/T1 disease) within 12 months of receiving adequate BCG (at least five of six doses doses of an initial induction course plus either at least two of three doses of maintenance therapy or at least two of six doses of a second induction course); or (b) Recurrent high-grade Ta/T1 disease within 6 months of completion of adequate BCG (at least five of six doses of an initial induction course plus either at least two of three doses of maintenance therapy or at least two of six doses of a second induction course); or (c) T1 high-grade disease at the first evaluation following an induction BCG course alone (at least five of six doses of an initial induction course).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Voluntary written informed consent and HIPAA authorization and agree to comply with all protocol-specified procedures and follow-up evaluations

Exclusion Criteria:

* Recurrence of BCG unresponsive Ta/T1 disease (without presence of CIS) > 6 months after last BCG instillation or BCG unresponsive CIS > 12 months after last BCG instillation.
* Life expectancy <2 years
* Any of the following clinical laboratory values at the time of enrollment: (1) Absolute neutrophil count (ANC) <800/µL or (2) Platelets < 50,000/µL
* Liver function abnormalities as indicated by ongoing hepatic enzyme elevation (AST or ALT) >2 times upper limit of normal (ULN)
* Renal insufficiency as indicated by a creatinine level >3 times ULN
* History of or evidence of muscle-invasive, locally advanced, metastatic and/or extravesical bladder cancer (inclusive of the prostatic urethra); or any other cancer within the past 5 years that is progressing or requires active treatment. Exceptions are adequately treated basal cell or squamous cell skin cancer that has undergone potentially curative therapy or in situ cervical cancer; and adequately treated stage I or II cancer or stable prostate cancer from which the patient is currently in complete remission, and is under active surveillance or hormone control.
* Symptomatic congestive heart failure (CHF), New York Heart Association (NYHA) Class III or IV heart failure or other clinical signs of severe cardiac dysfunction
* Severe/unstable angina pectoris, or myocardial infarction within 6 months prior to study entry
* History or evidence of uncontrollable central nervous system (CNS) disease
* Active systemic infection requiring parenteral antibiotic therapy. All prior infections must have resolved following optimal therapy
* Concurrent febrile illness, active urinary tract infection, active tuberculosis, a history of hypotension or anaphylactic reactions
* Ongoing chronic systemic steroid therapy required (>10 mg oral prednisone daily or equivalent)
* Women who are pregnant or nursing. Female patients of childbearing potential must have a negative pregnancy test and must adhere to using a medically acceptable method of birth control prior to screening and agree to continue its use during the study and for 30 days after the last dose of study drug, or be surgically sterilized (e.g., hysterectomy or tubal ligation). Women of childbearing potential are defined as any female who has experienced menarche and who is NOT permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause. Males must agree to use barrier methods of birth control while on study and for 90 days post last dose of study drug.
* Patients currently receiving investigational or commercial anti-cancer agents or anti-cancer therapies other than BCG, ALT-803 and supportive care therapies for active disease.
* Concurrent use of other investigational agents (not including FDA authorized drugs for the prevention and treatment of COVID-19).
* Other illness or condition, including laboratory abnormalities, which in the opinion of the Investigator would exclude the patient from participating in this study. This includes, but is not limited to, serious medical conditions or psychiatric illness likely to interfere with participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response | 60 Months
  Cohort A & Cohort C: Assess incidence of complete response of CIS (with or without Ta/T1 papillary disease) patients at any time
Disease-Free Rate | 12 Months
  Cohort B: Assess disease-free rate at 12 months since first study treatment

SECONDARY OUTCOMES:
Response | 60 months
  Cohort A & Cohort C: Assess duration of complete response Cohort B: Assess disease-free survival
Response | 6 months
  Cohort A & Cohort C: Assess complete response rate at 6 months. Cohort B: Assess disease-free rate at 6 months
Response | 9 months
  Cohort A & Cohort C: Assess complete response rate at 9 months. Cohort B: Assess disease-free rate at 9 months
Response | 12 months
  Cohort A & Cohort C: Assess complete response rate at 12 months. Cohort B: Assess disease-free rate at 12 months
Response | 18 months
  Cohort A & Cohort C: Assess complete response rate at 18 months. Cohort B: Assess disease-free rate at 18 months
Response | 24 months
  Cohort A & Cohort C: Assess complete response rate at 24 months. Cohort B: Assess disease-free rate at 24 months
Complete Response | 60 months
  Assess complete response rate at any time of CIS patients per central pathology review Duration of complete response (all recurrent bladder cancer, including low grade Ta disease)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Chamie, MD, Principal Investigator — University of California, Los Angeles
Locations (28):
- United States (28):
  - Alaska Clinical Research Center, Anchorage, Alaska
  - Arkansas Urology, Little Rock, Arkansas
  - UCLA Department of Urology, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Skyline Urology, Sherman Oaks, California
  - Skyline Urology, Torrance, California
  - Urology Associates, PC, Englewood, Colorado
  - University of Miami Miller School of Medicine-Sylvester Comprehensive Cancer Center, Miami, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Dwight D. Eisenhower Army Medical Center, Augusta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Adult & Pediatric Urology, Omaha, Nebraska
  - Accument Rx, Albuquerque, New Mexico
  - Roswell Park Cancer Insitute, Buffalo, New York
  - Winthrop University Hospital Department of Urology, Garden City, New York
  - Integrated Medical Professionals, New York, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Virginia Urology, Richmond, Virginia
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang SS, Chamie K, Kramolowsky E, Gonzalgo ML, Agarwal PK, Bassett JC, Bjurlin M, Cher ML, Clark W, Cowan BE, David R, Goldfischer E, Guru K, Jalkut MW, Kaffenberger SD, Kaminetsky J, Corcoran A, Koo AS, Sexton WJ, Tikhonenkov SN, Shah MS, Trabulsi EJ, Trainer AF, Spilman P, Huang M, Bhar P, Drusbosky LM, Sender L, Brown B, Reddy S, Soon-Shiong P. Prolonged Progression-Free Survival, Disease-Free Survival, and Cystectomy Avoidance With IL-15 Receptor Lymphocyte-Stimulating Agent NAI Plus Bacillus Calmette-Guerin in Bacillus Calmette-Guerin-Unresponsive Papillary-Only Nonmuscle-Invasive Bladder Cancer. J Urol. 2026 Jan;215(1):44-56. doi: 10.1097/JU.0000000000004782. Epub 2025 Sep 16. PMID 40956664
- [Derived] Chamie K, Chang SS, Rosser CJ, Kramolowski E, Gonzalgo ML, Sexton WJ, Spilman P, Sender L, Reddy S, Soon-Shiong P. N-803 Plus BCG Treatment for BCG-Naive or -Unresponsive Non-Muscle Invasive Bladder Cancer: A Plain Language Review. Future Oncol. 2024;20(31):2307-2317. doi: 10.1080/14796694.2024.2363744. Epub 2024 Jul 2. PMID 38953850